CLINICAL TRIAL: NCT03722355
Title: A Phase III Comparison of Hyperfractionated Radiation Therapy (RT) With BCNU and Conventional RT With BCNU for Supratentorial Malignant Glioma
Brief Title: Hyperfractionated RT With BCNU Versus Conventional RT With BCNU for Supratentorial Malignant Glioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 9006
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2018-10

CONDITIONS: Glioma; Glioblastoma Multiforme; Astrocytoma
Keywords: Glioma; Glioblastoma; Glioblastoma multiforme; Astrocytoma
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma | interventions — Carmustine; carmustine, poliferprosan 20 drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Conventional RT + Carmustine (Active Comparator): Conventional RT: 60.0 Gy/30 fractions/2.0 Gy once daily + carmustine 80 mg/m2 IV on Days 1, 2, 3 of RT then every 8 weeks for 6 cycles
  Interventions: Radiation: Conventional RT; Drug: Carmustine
- Arm 2: Hyperfractionated RT + Carmustine (Experimental): Hyperfractionated RT: 72.0 Gy/60 fractions/6 weeks/1.2 Gy BID + carmustine 80 mg/m2 IV on Days 1, 2, 3 of RT and then every 8 weeks for 6 cycles
  Interventions: Radiation: Hyperfractionated RT; Drug: Carmustine

INTERVENTIONS:
Radiation: Conventional RT — Radiation therapy
  Arms: Arm 1: Conventional RT + Carmustine
Radiation: Hyperfractionated RT — Radiation therapy
  Arms: Arm 2: Hyperfractionated RT + Carmustine
Drug: Carmustine — Chemotherapy
  Other Names: BCNU; Gliadel

SUMMARY:
Hyperfractionated radiation therapy (RT) to 72.0 Gy with BCNU will be compared to conventional radiation therapy to 60.0 Gy with BCNU to determine if hyperfractionated RT can improve the median survival time of adults with supratentorial malignant gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed glioblastoma multiforme (with areas of necrosis), malignant astrocytoma and astrocytoma with foci of anaplasia
* Karnofsky Performance Score ≥ 60
* Absolute Neutrophil count ≥ 1,500
* Platelets ≥ 100,000
* BUN ≤ 25
* Creatinine ≤ 1.5
* Bilirubin ≤ 2.0
* Hemoglobin ≥ 10 gm
* SGOT < 2 x upper limit of normal
* SGPT < 2 x upper limit of normal

Exclusion Criteria:

* No prior radiation to the head or neck area, chemotherapy or radiosensitizer
* No malignancy with the past five years except non-melanomatous skin cancer or carcinoma in-situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 1990-11-09 (Actual); Primary Completion 1994-03-15 (Actual); Study Completion 2002-10-18 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From randomization to the date of death or last follow up, assessed up to 131 months.
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Walter J Curran, Jr., MD, Principal Investigator — Radiation Therapy Oncology Group

REFERENCES:
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/